CLINICAL TRIAL: NCT06022692
Title: Water-filtered Infrared A Radiation Whole-body Hyperthermia Combined With Immune Checkpoint Inhibitor Therapy for Advanced Gastrointestinal Tumours: A Prospective Open-label Single-arm Phase 2 Study
Brief Title: Hyperthermia Combined With Immune Checkpoint Inhibitor Therapy for Advanced Gastrointestinal Tumours
Acronym: HEAIS001
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pengyuan Liu (Other)
Collaborators: Zhejiang Hospital (Other)
Responsible Party: Sponsor-Investigator, Pengyuan Liu, Research Secretary, Zhejiang Hospital
Organization: Zhejiang Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZhejiangH
Record Dates: First submitted 2023-08-18; First posted 2023-09-05 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-09

CONDITIONS: Gastrointestinal Tumor
Keywords: hyperthermia; immune checkpoint inhibitor
MeSH Terms: conditions — Digestive System Neoplasms; Hyperthermia | interventions — tislelizumab; Immune Checkpoint Inhibitors; spartalizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hyperthermia combined with immune checkpoint inhibitor group (Experimental): The patients were treated with whole-body hyperthermia on days 1 and 8 of each HIT cycle along with administration of tislelizumab 200 mg on day 2 (24 h after the hyperthermia at day 1).
  Interventions: Device: Water-filtered infrared A radiation whole-body hyperthermia (HECKEL 3000MT-4T, Germany); Drug: tislelizumab (BeiGene, China) combined with PD-1 inhibitor

INTERVENTIONS:
Device: Water-filtered infrared A radiation whole-body hyperthermia (HECKEL 3000MT-4T, Germany) — The patients were treated with whole-body hyperthermia (HECKEL 3000MT-4T, Germany)) on days 1 and 8 of each hyperthermia combined with immune checkpoint inhibitor treatment cycle along with administration of tislelizumab (BeiGene, China) 200 mg on day 2 (24 hours after the hyperthermia at day 1).
Drug: tislelizumab (BeiGene, China) combined with PD-1 inhibitor — The patients were treated with whole-body hyperthermia (HECKEL 3000MT-4T, Germany)) on days 1 and 8 of each hyperthermia combined with immune checkpoint inhibitor treatment cycle along with administration of tislelizumab (BeiGene, China) 200 mg on day 2 (24 hours after the hyperthermia at day 1).
  Other Names: Immune checkpoint inhibitor; PD-1 antibody

SUMMARY:
Gastrointestinal tumours (GITs) are the most common and fatal cancers worldwide; 96% of GITs show the microsatellite-stable (MSS)/proficient mismatch repair (pMMR) phenotype, and these tumours have a poor response to immune checkpoint inhibitor (ICI) therapy. Hyperthermia combined with ICI treatment (HIT) has been reported to show a synergistic sensitisation effect in numerous basic studies. This study aimed to validate the effectiveness, safety, and feasibility of water-filtered infrared A radiation (WIRA) whole-body hyperthermia combined with PD-1 inhibitor therapy and evaluate the real-world clinical application prospects of HIT. This open-label single-arm phase 2 clinical trial aimed to enrol advanced GIT patients with the MSS/pMMR phenotype in the East Asian population who had received third-line or higher treatment. The patients were treated with whole-body hyperthermia on days 1 and 8 of each HIT cycle along with administration of tislelizumab 200 mg on day 2 (24 h after the hyperthermia at day 1). The primary outcome was the disease control rate (DCR), while the secondary outcomes were progression-free survival (PFS), overall survival (OS), safety, and improvement in quality of life.

DETAILED DESCRIPTION:
The specific treatment process is shown in the trial flow diagram. The patients underwent WIRA whole-body hyperthermia on days 1 and 8 of each HIT cycle. On day 2 (24 h after hyperthermia on day 1), 200 mg of tislelizumab prepared with 100 mL of normal saline was intravenously administered for less than 30 min. After six HIT cycles, tislelizumab was administered intravenously every 21 days until drop-out. For quality control of hyperthermia, the core temperature was set to 38·5-39·5 °C and measured using a rectal temperature-sensing probe. Hyperthermia was considered to have been achieved when this temperature range was recached and maintained for 60 min. Each hyperthermia session lasted for 2 h, including a 30-min heating stage, a 60-min insulation stage, and a 30-min cooling stage. Clinical data were collected every two HIT treatment cycles and evaluated using the RECIST version 1.1 standard.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced GIT who have previously received third-line or above treatment.
* Patients are aged 18-75.
* Patients with at least one measurable tumor lesion.
* Patients' all physiological indexes meet the HIT requirements.

Exclusion Criteria:

* Patients have participated in other clinical trials within 4 weeks before enrollment.
* Patients contraindicate to whole-body hyperthermia.
* Patients contraindicate to immunotherapy.
* Patients cannot fully cooperate with HIT and follow-up.
* Pregnant or lactating women.
* Other circumstances may affect the results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
disease control rate (DCR) | up to 6 months
  DCR=(PR+CR) / (PD+SD+PR+CR) * 100%

SECONDARY OUTCOMES:
progression-free survival (PFS) | up to 36 months
  The time between enrollment and tumor progression (in any aspect) or death (for any reason).
overall survival (OS) | up to 36 months
  The time between enrollment and death (for any reason).

CONTACTS AND LOCATIONS:
Overall Officials: Jun Chen, Study Director — Zhejiang Hospital
Locations (1):
- Zhejiang Hospital, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No